CLINICAL TRIAL: NCT03989414
Title: A Phase 1/2, Multicenter, Open-label, Study to Determine the Recommended Dose and Regimen, and Evaluate the Safety and Preliminary Efficacy of CC-92480 in Combination With Standard Treatments in Subjects With Relapsed or Refractory Multiple Myeloma (RRMM) and Newly Diagnosed Multiple Myeloma (NDMM)
Brief Title: A Study to Determine the Recommended Dose and Regimen and to Evaluate the Safety and Preliminary Efficacy of CC-92480 in Combination With Standard Treatments in Participants With Relapsed or Refractory Multiple Myeloma (RRMM) and Newly Diagnosed Multiple Myeloma (NDMM)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-92480-MM-002; U1111-1233-5619 (Other: WHO); 2023-505219-19 (Registry Identifier: EU CT number)
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma
Keywords: Relapsed or Refractory Multiple Myeloma; Newly Diagnosed Multiple Myeloma; Multiple Myeloma; CC-92480
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bortezomib; Dexamethasone; daratumumab; carfilzomib; elotuzumab; isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Cohort A: CC-92480 with bortezomib and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Bortezomib; Drug: Dexamethasone
- Cohort C: CC-92480 with carfilzomib and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Dexamethasone; Drug: Carfilzomib
- Cohort H: CC-92480 with elotuzumab and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Dexamethasone; Drug: Elotuzumab
- Cohort I: CC-92480 with isatuximab and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Dexamethasone; Drug: Isatuximab
- Cohort D: CC-92480 with bortezomib and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Bortezomib; Drug: Dexamethasone
- Cohort F: CC-92480 with carfilzomib and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Dexamethasone; Drug: Carfilzomib
- Cohort J: CC-92480 with elotuzumab and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Dexamethasone; Drug: Elotuzumab
- Cohort K: CC-92480 with isatuximab and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Dexamethasone; Drug: Isatuximab
- Cohort G: CC-92480 with bortezomib and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Bortezomib; Drug: Dexamethasone
- Subcohort B1: CC-92480 with daratumumab and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Dexamethasone; Drug: Daratumumab
- Subcohort B2: CC-92480 with daratumumab and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Dexamethasone; Drug: Daratumumab
- Subcohort B3: CC-92480 with daratumumab and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Dexamethasone; Drug: Daratumumab
- Subcohort E1: CC-92480 with daratumumab and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Dexamethasone; Drug: Daratumumab
- Subcohort E2: CC-92480 with daratumumab and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Dexamethasone; Drug: Daratumumab
- Subcohort E3: CC-92480 with daratumumab and dexamethasone (Experimental)
  Interventions: Drug: CC-92480; Drug: Dexamethasone; Drug: Daratumumab

INTERVENTIONS:
Drug: CC-92480 — Specified dose on specified days
  Other Names: BMS-986348; mezigdomide
Drug: Bortezomib — Specified dose on specified days
  Arms: Cohort A: CC-92480 with bortezomib and dexamethasone; Cohort D: CC-92480 with bortezomib and dexamethasone; Cohort G: CC-92480 with bortezomib and dexamethasone
Drug: Dexamethasone — Specified dose on specified days
Drug: Daratumumab — Specified dose on specified days
  Arms: Subcohort B1: CC-92480 with daratumumab and dexamethasone; Subcohort B2: CC-92480 with daratumumab and dexamethasone; Subcohort B3: CC-92480 with daratumumab and dexamethasone; Subcohort E1: CC-92480 with daratumumab and dexamethasone; Subcohort E2: CC-92480 with daratumumab and dexamethasone; Subcohort E3: CC-92480 with daratumumab and dexamethasone
Drug: Carfilzomib — Specified dose on specified days
  Arms: Cohort C: CC-92480 with carfilzomib and dexamethasone
Drug: Elotuzumab — Specified dose on specified days
  Arms: Cohort H: CC-92480 with elotuzumab and dexamethasone; Cohort J: CC-92480 with elotuzumab and dexamethasone
Drug: Isatuximab — Specified dose on specified days
  Arms: Cohort I: CC-92480 with isatuximab and dexamethasone; Cohort K: CC-92480 with isatuximab and dexamethasone
Drug: Carfilzomib — Specified dose on specified days
  Arms: Cohort F: CC-92480 with carfilzomib and dexamethasone

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of CC-92480 in combination with standard treatments.

ELIGIBILITY:
Inclusion Criteria:

• Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2

For participants in Cohorts A, B, C, D, E, F, H, I, J, and K the following inclusions will also apply:

* Documented diagnosis of multiple myeloma (MM) and measurable disease
* Documented disease progression during or after their last antimyeloma regimen
* Achieved a response (minimal response [MR] or better) to at least 1 prior treatment regimen

Exclusion Criteria:

* Plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or clinically significant amyloidosis
* Known central nervous system (CNS) involvement with myeloma
* Received immunosuppressive medication within the last 14 days of initiating study treatment
* Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Recommended Dose | Up to approximately 3 years
Recommended regimen as measured by dose-limiting toxicities | Up to approximately 3 years
Number of participants with Adverse Events (AEs) | From first participant first visit until 28 days after the last subject discontinues study treatment, up to 5 years
Overall response rate (ORR) | Up to approximately 5 years

SECONDARY OUTCOMES:
Time-to-response (TTR) | Up to approximately 5 years
Duration of response (DOR) | Up to approximately 5 years
Complete Response (CR) rate | Up to approximately 5 years
Very good partial response (VGPR) rate - Cohorts D and E | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (49):
- United States (16):
  - Local Institution - 119, Denver, Colorado
  - Local Institution - 104, Tampa, Florida
  - Local Institution - 108, Atlanta, Georgia
  - Local Institution - 112, Chicago, Illinois
  - Local Institution - 107, Chicago, Illinois
  - Local Institution - 117, Boston, Massachusetts
  - Local Institution - 101, Boston, Massachusetts
  - Local Institution - 118, Boston, Massachusetts
  - Local Institution - 113, Detroit, Michigan
  - Local Institution - 106, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Local Institution - 110, Winston-Salem, North Carolina
  - Local Institution - 115, Columbus, Ohio
  - Local Institution - 114, Nashville, Tennessee
  - Local Institution - 116, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Canada (5):
  - Local Institution - 201, Calgary, Alberta
  - Local Institution - 205, Edmonton, Alberta
  - Local Institution - 204, Halifax, Nova Scotia
  - Local Institution - 203, Toronto, Ontario
  - Local Institution - 202, Montreal, Quebec
- Czechia (3):
  - Local Institution - 802, Brno
  - Local Institution - 801, Ostrava-Poruba
  - Local Institution - 803, Prague
- Denmark (2):
  - Local Institution - 902, Odense
  - Local Institution - 903, Vejle
- France (5):
  - Local Institution - 703, Lille
  - Local Institution - 705, Marseille
  - Local Institution - 704, Nantes
  - Local Institution - 701, Toulouse
  - Local Institution - 702, Tours
- Germany (5):
  - Local Institution - 604, Freiburg im Breisgau
  - Local Institution - 605, Hamburg
  - Local Institution - 601, Heidelberg
  - Local Institution - 602, München
  - Local Institution - 603, Würzburg
- Local Institution - 301, Athens, Greece
- Italy (4):
  - Local Institution - 404, Brescia
  - Local Institution - 401, Milan
  - Local Institution - 403, Reggio Emilia
  - Local Institution - 402, Torino
- Spain (8):
  - Local Institution - 504, Badalona
  - Local Institution - 508, Madrid
  - Local Institution - 501, Madrid
  - Local Institution - 506, Málaga
  - Local Institution - 505, Pamplona
  - Local Institution - 502, Salamanca
  - Local Institution - 503, Santander
  - Local Institution - 507, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT03989414.html